CLINICAL TRIAL: NCT04793269
Title: Long COVID Syndrom: Charakterisierung Eines Neuen Krankheitsbildes
Brief Title: Characteristics of Long COVID-19 Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Christian Clarenbach (Other)
Responsible Party: Sponsor-Investigator, Christian Clarenbach, Sponsor Investigator, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2021-00280
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Long COVID Syndrome
Keywords: long COVID; post COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Long COVID: Patients with long COVID syndrome
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
Characterization of patients with long COVID syndrome including symptoms, medical history and persistent organ damage.

DETAILED DESCRIPTION:
Some people are very hesitant to recover from a COVID-19 infection and present persistent symptoms. The participants still suffer after the acute phase of the infection from shortness of breath, coughing, chest pain or fatigue. Therefore, a special interdisciplinary consultation was built. The consulatation is not only addressed to people who have been hospitalized due to COVID-19, but also to those with mild symptoms during infection. During the consultation hours, personal health data are collected that serves as the basis for this research project.

ELIGIBILITY:
Inclusion Criteria:

* Long COVID syndrome
* age >= 18 years
* Informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with long COVID syndrome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dyspnea | once through study completion, an average of 6 months.
  modified medical research council (scale from 0 to 4). The higher the score the worse the symptoms.
self-addressed Quality of life | once through study completion, an average of 6 months
  Short form health 36 questionnaire with 8 domains, each rated from 0-100. The higher the score the better subjective quality of life.
Thoracic pain | once through study completion, an average of 6 months
  assessed by medical interview (reported as yes or no)
Medical history | once through study completion, an average of 6 months
  List of relevant morbidities assessed as present/not present by medical interview (e.g. respiratory, cardial, neurological, psychiatric diseases by interview and medical records)
Fibrosis | once through study completion, an average of 6 months
  Assessed by chest CT, rated as present/not present
Myocardial damage | once through study completion, an average of 6 months
  Assessed by myocardial damage, rated as present/not present

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Clarenbach, MD, Study Chair — University Hospital Zurich, Pulmonology
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD will be shared on request

REFERENCES:
- [Derived] Malesevic S, Sievi NA, Baumgartner P, Roser K, Sommer G, Schmidt D, Vallelian F, Jelcic I, Clarenbach CF, Kohler M. Impaired health-related quality of life in long-COVID syndrome after mild to moderate COVID-19. Sci Rep. 2023 May 12;13(1):7717. doi: 10.1038/s41598-023-34678-8. PMID 37173355